CLINICAL TRIAL: NCT05801640
Title: Facilitated Tucking Position and Reiki Efficacy in Orogastric Tube Insertion in Preterm Infants: Randomized Controlled Trial
Brief Title: Facilitated Tucking Position and Reiki Efficacy in Orogastric Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Küçükoğlu (Other)
Responsible Party: Sponsor-Investigator, Sibel Küçükoğlu, Professor Ph.D., Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SelcukH01
Record Dates: First submitted 2022-10-26; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Premature; Feeding Behavior; Infant, Premature, Diseases
Keywords: Premature; Reiki; Pain; Facilitated tucking
MeSH Terms: conditions — Premature Birth; Feeding Behavior; Infant, Premature, Diseases; Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Parallel Assignment After explaining the study to eligible and accepting parents, informed consent signatures will be obtained. Randomization will be done after obtaining informed consent from the parent. Random assignment will be made to one control group or one intervention group (faciliated tucking position:1, reiki: 1) with sequentially numbered, sealed, opaque envelopes containing randomly generated numbers in randomization. These envelopes are for a person not involved in any other trial procedure. Will be made by Randomization will be performed using the random numbers table.
Who Masked: Participant, Outcomes Assessor
Masking Description: Single (participant and outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Faciliated tucking position (Experimental): Experiment group will receive faciliated tucking position throughout the OG inserting. The faciliated tucking position will be applied 3 minutes before the orogastric (OG) tube is inserted. This intervention will be applied throughout the OG inserting process. The application will continue for 3 more minutes after the OG is inserted.
  Interventions: Other: Facilitated Tucking Position
- Reiki (Experimental): Experiment group will receive reiki throughout the OG inserting. This group will be take reiki 3 minutes before the orogastric (OG) tube is inserted. This intervention will be applied throughout the OG inserting process. The intervention will continue for 3 more minutes after the OG is inserted.
  Interventions: Other: Reiki
- Control Group (No Intervention): The routine OG insertion procedure of the clinic will be performed for the control group infants without any intervention. The group will received no further intervention.

INTERVENTIONS:
Other: Facilitated Tucking Position — The fetal position was given by the researcher. In the fetal position, the lower and upper extremities of the baby were kept in the flexed position by hand and placed in the side-lying position close to the midline.
  Arms: Faciliated tucking position
Other: Reiki — Reiki was applied to areas called chakras (forehead, throat, heart, stomach, feet and hands). A total of 15 minutes were applied in the form of 12 minutes touches in each chakra region.
  Arms: Reiki

SUMMARY:
The aim of this study is to determine the effects of faciliated tucking and reiki given manually during orogastric tube insertion in preterm infants treated in the NICU on stress, pain and physiological parameter (heartbeat, blood pressure, SpO2 and respiratory rate) levels.

DETAILED DESCRIPTION:
Regardless of the severity and duration, preterm infants give physiological and behavioral responses to a painful application. While infants show behavioral responses such as crying, changes in facial expressions, acceleration or deceleration in motor movements during painful interventions, they may subjectively show changes in physiological parameters such as heart rate, respiratory rate, blood pressure, and decrease in saturation value. Because preterm infants are sensitive to many stress factors and due to reasons such as separation from the mother during the treatment process, environments with excessive light, sound and temperature changes, and the absence of a single caregiver. They do not yet have the physiological maturity to cope with painful interventions. This randomized controlled trial was planned to determine the changes in stress, pain, and physiological parameters of faciliated tucking and reiki administered during orogastric tube insertion in preterm infants 32-37 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* 32-37 Gestational weeks,
* From the postnatal 3rd day,
* Feeding with orogastric tube
* Apgar >5

Exclusion Criteria:

* Premature infants with congenital anomaly, malformation
* Premature infants on mechanical ventilator
* Premature infants receiving sedation

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Newborn Information Form | One measurement- Half an hour before the intervention
  The descriptive characteristics form was based on a literature review conducted by the researcher (Axelin, Salanterä & Lehtonen, 2006; Kucukoglu, Kurt & Aytekin, 2015; Yin, Yang, Lee, Li, Hua & Liaw, 2015). The form consisted of items on gestational age, postnatal age, gender, birth weight (grams), type of delivery, 1st and 5th minute Apgar score, etc.
Neonatal Stress Scale | First measurement- 1 minute before OG tube insertion
  To determine the effect of facilitated tucking position on stress score during OG procedure in preterm infants.
  It was developed by Ceylan and Bolışık (2017) to evaluate the stress level in premature infants. The scale is suitable for use by nurses. The scale includes 8 subgroups including facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities and posture, and consists of a total of 24 items in 3-likert type. In scoring, each subgroup is evaluated between 0-2 points. The score obtained from the scale is a minimum of 0 points and a maximum of 16 points. This form filled by a clinical nurse and researcher 2 times before, and after the procedure.
Neonatal Stress Scale | Second measurement- 1 minute after OG tube insertion
  To determine the effect of facilitated tucking position on stress score during OG procedure in preterm infants.
  It was developed by Ceylan and Bolışık (2017) to evaluate the stress level in premature infants. The scale is suitable for use by nurses. The scale includes 8 subgroups including facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities and posture, and consists of a total of 24 items in 3-likert type. In scoring, each subgroup is evaluated between 0-2 points. The score obtained from the scale is a minimum of 0 points and a maximum of 16 points. This form filled by a clinical nurse and researcher 2 times before, and after the procedure.
Physiological Parameter Tracking Chart | First measurement- 1 minute before OG tube insertion
  It is a form that includes the heart rate, oxygen saturation value and respiratory rate. This form filled by a clinical nurse 2 times before and after the procedure, by a clinical nurse other than the person performing the research.
Physiological Parameter Tracking Chart | Second measurement 1 minute after OG tube insertion
  It is a form that includes the heart rate, oxygen saturation value and respiratory rate. This form filled by a clinical nurse 2 times before and after the procedure, by a clinical nurse other than the person performing the research.
The premature infant pain profile-revised (PIPP-R) | Two measurements: First measurement- 1 minute before OG tube insertion
  The PIPP-R scale includes 3 behavioral (fringing, squeezing eyes, nasolobial-groove), 2 physiological (heart rate and oxygen saturation) and 2 contextual (behavioral status and gestational age) items used in the assessment of pain in newborns.This form filled by a clinical nurse and researcher 2 times before, and after the procedure. The PIPP-R is a Likert-type scale. In scoring the scale, items related to physiological and behavioral parameters are scored as 0,1,2,3 for each variable, reflecting the difference between the initial state and the values during the procedure.
The premature infant pain profile-revised (PIPP-R) | Second measurement 1 minute after OG tube insertion
  The PIPP-R scale includes 3 behavioral (fringing, squeezing eyes, nasolobial-groove), 2 physiological (heart rate and oxygen saturation) and 2 contextual (behavioral status and gestational age) items used in the assessment of pain in newborns.This form filled by a clinical nurse and researcher 2 times before, and after the procedure. The PIPP-R is a Likert-type scale. In scoring the scale, items related to physiological and behavioral parameters are scored as 0,1,2,3 for each variable, reflecting the difference between the initial state and the values during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Onal, M.Sc., Principal Investigator — Nigde Omer Halisdemir University; Halil Degirmencioglu, Medicine, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Kucukoglu S, Kurt S, Aytekin A. The effect of the facilitated tucking position in reducing vaccination-induced pain in newborns. Ital J Pediatr. 2015 Aug 21;41:61. doi: 10.1186/s13052-015-0168-9. PMID 26293573
- [Result] Im H, Kim E. Effect of Yakson and Gentle Human Touch versus usual care on urine stress hormones and behaviors in preterm infants: a quasi-experimental study. Int J Nurs Stud. 2009 Apr;46(4):450-8. doi: 10.1016/j.ijnurstu.2008.01.009. Epub 2008 Mar 18. PMID 18353332